CLINICAL TRIAL: NCT02982902
Title: Antigen Specific Adoptive T Cell Therapy for Opportunistic Cytomegalovirus Infection Occurring After Stem Cell Transplant
Brief Title: T Cell Therapy of Opportunistic Cytomegalovirus Infection
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mari Dallas (Other)
Responsible Party: Sponsor-Investigator, Mari Dallas, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE1Z16
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2025-10-22 (Actual); Status verified 2025-09

CONDITIONS: Cytomegalovirus Infections; Hematopoietic Stem Cell Transplant; Opportunistic Infections
Keywords: Immunotherapy; T-Cell Therapy; Lymphoproliferative Disorder
MeSH Terms: conditions — Cytomegalovirus Infections; Opportunistic Infections; Lymphoproliferative Disorders | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CMV specific adoptive t-cells (Experimental): This study involves a one-time infusion of the experimental CMV specific adoptive t-cells. After this infusion, patients will be followed for 4 weeks.
  Interventions: Biological: CMV specific adoptive t-cells

INTERVENTIONS:
Biological: CMV specific adoptive t-cells — It is expected that the cell dose will be in the range of 10^3 - 10^5 virus - specific, antigen selected T cells per kg of recipient weight.
  Other Names: immunotherapy

SUMMARY:
The purpose of this study is to determine if a specific type of cell-based immunotherapy, using T-cells from a donor that are specific against cytomegalovirus (CMV) is feasible to treat infections by CMV.

Adoptive T-cell therapy is an investigational (experimental) therapy that works by using the blood of a donor and selecting the T-cells that can respond against a specific infectious entity. These selected T-cells are then infused to the patient, to try to give the immune system the ability to fight the infection. Adoptive T-cell therapy is experimental because it is not approved by the Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
The primary objective of this study is to determine the feasibility of the treatment of opportunistic cytomegalovirus (CMV) infections after hematopoietic stem cell transplant (HSCT) with virus-specific, antigen-selected T-cells, selected using the CliniMACS prodigy system.

Secondary Objective(s)

* To describe the safety profile of the infusion of CMV- specific, antigen selected T-cells.
* To describe the toxicities related to infusion of CMV- specific, antigen selected T-cells.
* To describe the rate of eradication of opportunistic CMV infections after HSCT and and treatment with CMV-specific, antigen-selected T-cells using the CliniMACS Prodigy System.

This feasibility study will include a single treatment cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have received allogeneic hematopoietic stem cell transplant and be greater than 30 days post-transplant at the time of registration
* Patients must have documented opportunistic CMV infection, or reactivation; the criteria include (both of the following criteria must be met)

  * Patients may have asymptomatic viremia (>1000 copies/ml) OR presence of symptoms secondary to CMV infection, AND
  * Patients must have ONE OF THE NEXT FOUR CRITERIA:

    * Absence of an improvement of viral load after ≥ 14 days of antiviral therapy with ganciclovir, valganciclovir or foscarnet (decrease by at least 1 log, i.e. 10-fold) or
    * New, persistent and/or worsening CMV-related symptoms, signs and/or markers of end organ compromise while on antiviral therapy with ganciclovir, valganciclovir or foscarnet, or
    * Have contraindications or experience adverse effects of antiviral therapy with ganciclovir, valganciclovir or foscarnet.
    * Second recurrence of CMV viremia, CMV-related symptoms, signs and/or markers of end organ compromise.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 3
* Women of child-bearing potential and men must agree to use adequate contraception (double barrier method of birth control or abstinence) 4 weeks prior to study entry, for the duration of study participation and for 3 months after completing treatment.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document, or assent document.

Exclusion Criteria:

* Pregnant or breastfeeding women are excluded from this study.
* Patients with opportunistic viral infections other than CMV.
* Patients with active, grade 2-4, acute graft vs. host disease (GVHD), chronic GVHD or any condition requiring high doses of glucocorticosteroid (>0.5 mg/kg/day prednisone or its equivalent) as treatment
* Treatment with antithymocyte globulin within 28 days of planned infusion of virus - specific, antigen selected T cells.
* Treatment with virus - specific T cells within 6 weeks (42 days) of planned infusion.

Donor eligibility

* Related donor of T cells must be at least partially HLA compatible, matching with recipient in at least 3/6 HLA loci (HLA-A, HLA-B, and HLA-DRB1 loci will be considered for this).
* Must have evidence of a serologic response (i.e. be seropositive) against CMV.
* Age ≥ 18 years
* Must meet the criteria for donor selection defined in the Standard Operating Procedures of University Hospitals Seidman Cancer Center Stem Cell Transplant Program
* Must be capable of undergoing a single standard 2 blood volume leukapheresis or donation of one unit of whole blood

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-27 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 100 days after transplant
  To determine the feasibility of the intervention, the study will record the incidence of adverse events, including graft versus host disease and other complications will be evaluated using binomial distribution theory and their 95% confidence intervals (CIs) will be also estimated using Wilson's method

SECONDARY OUTCOMES:
Eradication rate of opportunistic CMV infections | Up to 100 days after transplant
  The eradication rate will be the disappearance of opportunistic CMV infections with the use of CMV-specific, antigen-selected T cells using the CliniMACS Prodigy System over the total number CMV infections.
response rate | Up to 100 days after transplant
  A response rate of 25% is considered unacceptable; and the anticipated response rate is approximately 55% for the study population using the cell therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mari H Dallas, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No